CLINICAL TRIAL: NCT05444725
Title: Investigating Barriers for Decision Making in a Danish Breast Cancer Screening Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-051-000001, 2563
Record Dates: First submitted 2022-06-03; First posted 2022-07-06 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer Female; Mammography Screening; Decision Making; Information Seeking Behavior
MeSH Terms: conditions — Information Seeking Behavior

STUDY DESIGN:
Intervention Model Description: Self administered questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage of decision making (Other): Same questionnaire for all three arms except validated question "Stage of decision making" followed by question about participation in screening or not when invited at age 50.
  This is not an intervention but a survey study with three different versions of the questionnaire.
  Interventions: Other: Stage of Decision Making
- Choice framing (Other): Same questionnaire for all three arms except text and question presenting breast cancer screening as a choice (between screening and alternative of no screening) followed by question about participation in screening or not when invited at age 50.
  This is not an intervention but a survey study with three different versions of the questionnaire.
  Interventions: Other: Choice framing
- Opportunity framing (Other): Same questionnaire for all three arms except text and question presenting breast cancer screening as an opportunity (no presentation of alternative) followed by question about participation in screening or not when invited at age 50.
  This is not an intervention but a survey study with three different versions of the questionnaire.
  Interventions: Other: Opportunity Framing

INTERVENTIONS:
Other: Stage of Decision Making — Investigating preferences and attitudes towards breast cancer screening information, invitation, and decision making as well as barriers for breast cancer decision making. This will be done by using different framing of information (choice framing vs. opportunity framing), question about stage of decision making, and general questions about screening information and invitation.
  Arms: Stage of decision making
Other: Choice framing — Investigating preferences and attitudes towards breast cancer screening information, invitation, and decision making as well as barriers for breast cancer decision making. This will be done by using different framing of information (choice framing vs. opportunity framing), question about stage of decision making, and general questions about screening information and invitation.
  Arms: Choice framing
Other: Opportunity Framing — Investigating preferences and attitudes towards breast cancer screening information, invitation, and decision making as well as barriers for breast cancer decision making. This will be done by using different framing of information (choice framing vs. opportunity framing), question about stage of decision making, and general questions about screening information and invitation.
  Arms: Opportunity framing

SUMMARY:
The aim is to investigate potential barriers to informed decision making in a breast cancer screening context. This is a necessary step prior to developing and investigating improved information or decision aids in a Danish breast cancer screening context.

DETAILED DESCRIPTION:
In this study, preferences and attitudes towards breast cancer screening, invitation, and decision making among Danish women will be investigated. The aim is to gain knowledge about barriers for (informed) decision making in a Danish breast cancer screening context. The study will be conducted by sending out an online questionnaire to women aged 44-49 in Denmark. The questionnaire will be sent out using the official digital mail system, e-Boks, with an invitation, link, and login information to access the online questionnaire. The questionnaire will consist of background questions about the participants, questions related to the current information material and invitation to the Danish breast cancer screening program, and questions about decision making and informed choice. Women will be randomized to one of three questionnaires: 1) Questionnaire with "Stage of Decision Making" to investigate women's decision making process regarding participation in screening, 2) Questionnaire with choice framing (presentation of a choice between participation in breast cancer screening or no screening), or 3) Questionnaire with opportunity framing (only presentation of screening, no alternative) to investigate decision making process and impact of different framing. The main hypothesis for this study is that 80% of Danish women have already made their decision about screening participation when presented to the opportunity framing and 70% when presented to the choice framing.

1000 women will be invited to each group in this study and thus 3000 in total, as this is the minimum number satisfying the requirements for both the main hypothesis and secondary aims (not described in detail here). No similar studies were found, therefore, this sample size calculation is based on proportions of 50% to have enough power in our study. With a desired standard error no larger than 2.5%, 400 women are required (SE of a binomial random variable). Assuming 40% participation, a study population of 1000 women in each group is required.

Next, questionnaire data will be linked to register data on sociodemographic factors from Statistics Denmark.

The study is registered at Aarhus University's internal records: 2016-051-000001, 2563.

ELIGIBILITY:
Inclusion Criteria:

* All women living in Denmark in this age group

Exclusion Criteria:

* None

Ages: 44 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3000 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of women who have made the decision about screening participation prior to screening invitation. | The outcome is assessed when women answer the questionnaire sent out in late June 2022. It will take 5-10 minutes to answer the questionnaire. The questionnaire will be closed after 1.5-2 months.
  The main hypothesis for this study is that 80% of Danish women have already made their decision about screening participation when presented to the opportunity framing and 70% when presented to the choice framing. Further, a question about being more or less willing to participate after reading screening information will also provide information for this hypothesis.

SECONDARY OUTCOMES:
Prevalence of women not taking the presented screening information into account when making their decision about participation. | The outcome is assessed when women answer the questionnaire sent out in late June 2022. It will take 5-10 minutes to answer the questionnaire. The questionnaire will be closed after 1.5-2 months.
  This will be investigated by comparing the choice vs. opportunity framing, with questions about reading health information in general and about having read the information about breast cancer screening in this questionnaire. In addition, this will be investigated with questions about being more or less positive/negative about screening and more or less willing to participate after reading the screening information.
Prevalence of women not thinking of the screening participation as an actual (individual) choice but something to comply with when invited. | The outcome is assessed when women answer the questionnaire sent out in late June 2022. It will take 5-10 minutes to answer the questionnaire. The questionnaire will be closed after 1.5-2 months.
  This will be investigated using two statements about seeing the participation as an individual choice or as a recommendation from health authorities to comply with.
Prevalence of women not wanting to make an informed decision about their own health (and be responsible for their own health). | The outcome is assessed when women answer the questionnaire sent out in late June 2022. It will take 5-10 minutes to answer the questionnaire. The questionnaire will be closed after 1.5-2 months.
  This will be investigated with different statements about preferences regarding who should make the screening decision (the individual women or health authorities).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health, Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Not allowed by authorities.

REFERENCES:
- [Derived] Rossell EL, Bekker HL, Schonberg MA, Sonbo Kristiansen I, Borgquist S, Stovring H. Danish Women Make Decisions about Participation in Breast Cancer Screening prior to Invitation Information: An Online Survey Using Experimental Methods. Med Decis Making. 2024 Aug;44(6):674-688. doi: 10.1177/0272989X241248142. Epub 2024 May 4. PMID 38703097

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT05444725/SAP_000.pdf